CLINICAL TRIAL: NCT03935880
Title: Treatment of Hallux Rigidus With Synthetic Hemiarthroplasty Versus Cheilectomy: A Randomized Controlled Trial
Brief Title: Surgical Treatment for Great Toe Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty meeting recruitment goals
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1546; A536110 (Other: UW Madison); SMPH/ORTHO&REHAB/ORTHO (Other: UW Madison)
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cartiva Hemiarthroplasty (Active Comparator): Cartiva implant
  Interventions: Device: Cartiva Implant
- Cheilectomy (Active Comparator): Bone spur removal
  Interventions: Procedure: Cheilectomy

INTERVENTIONS:
Device: Cartiva Implant — Cartiva hemiarthroplasty: The procedure starts with a small incision over the top of the 1st MTP joint. The joint is exposed. Bone spurs on the metatarsal and proximal phalanx are resected, leaving approximately 2 mm of surrounding bone on the metatarsal head. A guide pin is placed within the metatarsal and a drill is then used to create a site for the implant. The implant is then placed using the implant introducer. The incision is then closed and a sterile dressing is placed.
  Arms: Cartiva Hemiarthroplasty
Procedure: Cheilectomy — Cheilectomy: A small incision is made over the top of the 1st MTP joint. The joint is exposed. Bone spurs on the metatarsal and proximal phalanx are resected. The top of the metatarsal head is then cut with a sagittal saw. Additional bone spurs are resected. The incision is closed and a sterile dressing is placed.
  Arms: Cheilectomy

SUMMARY:
After potential subjects determine that they would like surgical treatment of their great toe arthritis, study staff will approach them about the study. If subject decides to participate, they will be asked to fill out an informed consent. After the informed consent has been signed, study staff will collect subject demographics and medical/surgical history. The subject will be randomized into one of two surgical treatment options: cheilectomy or Cartiva hemiarthroplasty. The randomization ratio will be 1:1 and to ensure this randomization ratio, each randomization block will have 4-6 patients. After the surgery, the subject will have follow up visits at 2 weeks, 6 weeks, 3 months, 1 year, and 2 years post surgery. At these follow up visits, subjects will have a physical exam conducted, have their medical imaging reviewed, and fill out a data collection form which will include questionnaires and adverse event forms (when applicable). All of the above will apply to the 2 week visit, except for the administration of questionnaires/surveys. Additionally, subjects will have incision check, suture removal, and a physical completed during this visit.All study procedures for this study are considered standard of care. Patients would have these completed regardless of participation in the study.

DETAILED DESCRIPTION:
Hallux Rigidus is a common disorder that affects an estimated 1 in 40 people over the age of 50.4 While debate remains about the primary cause of this disorder, it is likely multifactorial with contributing factors including previous trauma, malalignment and underlying genetic influences.5 Regardless of the cause, the disorder can become progressive and significantly impact a patient's quality of life. Common symptoms include pain, swelling and limited range of motion. Patients often present with pain dorsally over the first metatarsophalangeal (MTP) joint secondary to osteophyte formation and swelling. This can restrict range of motion at this joint, as well as make daily activities, such as wearing closed-toed shoes, quite difficult.6 Furthermore, continued pain can lead to gait abnormalities with more weight bearing through the lateral aspect of the foot and potential transfer metatarsalgia.7

Along with physical exam to identify first MTP range of motion, joint swelling, erythema and palpable osteophyte formation, radiographic evaluation is part of the standard of care in hallux rigidus evaluation. Coughlin and Shurnas proposed a grading system that has become widely used, based on the radiographic findings and range of motion at the MTP joint.8 The grading system allowed clinicians to characterize patients from grade 0-4, helping guide treatment decisions.

Initial treatment is centered on pain relief with non-operative modalities. Modified shoe wear, custom orthotics with a Morton extension and activity modifications have all been shown to improve symptoms in some patients.7 For patients that fail non-operative therapies, a wide array of surgical options exist. For patients with Grade 1 and 2 hallux rigidus, joint sparing procedures have been primarily used, with the most common procedure being Cheilectomy. The Cheilectomy procedure involves removal of the dorsal osteophytes and 20-30% of the dorsal metatarsal head.3 The benefits of this procedure include the ability to improve joint mobility, while still leaving the potential for future fusion. Success rates have been reported between 72% and 100% in patients with grade 1 and 2 hallux rigidus.7 Controversy remains regarding cheilectomy in patients with grade 3 hallux rigidus however. Nicolosi et al found an average satisfaction rate of 85% in patients with grade 3 disease undergoing cheilectomy3. Additional studies, however have suggested high failure and revision rates in patients with grade 3 hallux rigidus.3

Joint fusion has become common place in the treatment of advanced stage hallux rigidus, including grade 3 and 4. High fusion rates and patient satisfaction has been proven with fusion procedures in the first MTP joint.7 However, the loss of motion at the first MTP joint associated with the fusion procedure can interfere with activities such as running and jumping, and can make shoe wear choices difficult2. These limitations led to the push for development of a joint replacement procedure, allowing for pain control and continued motion.

The use of silicone-based joint replacement has been met with mixed results, however concerns over the durability leading to implant fracture, osteolysis and difficulty of revision procedures has ultimately limited its use.9 Ceramic implants were found to have good short-term results, however concerns remain regarding the large amount of subsidence seen in follow up, as well as potential osteolysis10. Furthermore, the amount of bone stock remaining following this procedure could make revision procedures quite challenging. Given these mixed results, there remained a significant drive to identify a joint replacement-type procedure with a device that could maintain adequate bone stock, preserve motion and withstand the daily stresses the first MTP joint faces.

This led to the use of the Cartiva implant, a polyvinyl alcohol hydrogel implant. Following extensive safety and wear testing, it was determined that this implant would be well suited for use in patients with hallux rigidus. Indicated for grade 2, 3 and 4 hallux rigidus, the initial study of Cartiva effectiveness compared outcomes of the implant versus arthrodesis. The prospective, randomized control trial evaluated 202 patients, with over 2/3 undergoing the Cartiva procedure.2 Both short and midterm outcomes were very promising. 5-year revision rates were found to be 5% with no evidence of implant loosening or surrounding bone complication.11 Additionally, the Cartiva implant was found to be equivalent to the gold standard, arthrodesis, when it came to post-operative patient outcome scores, range of motion and complications.2

With promising results from initial clinical trials, further evaluation into the efficacy and indications for Cartiva is necessary. To date, there is no published literature comparing Cheilectomy to Cartiva. Both procedures have shown to have beneficial results in patients with grade 2 hallux rigidus, yet it is unclear if one procedure would be preferred in this population or certain subsets of patients. With an estimated revision rate around 9% following Cheilectomy, it is possible that Cartiva could decrease the need for additional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade 2 hallux rigidus using the grading system described by Coughlin and Shurnas.8
* Patients older than 18 and less than 88 years of age
* Patients will have the ability to perform the questionnaires and will complete the informed consent process.

Exclusion Criteria:

* Patients with the diagnosis of gout or inflammatory arthropathy
* Patients with inadequate bone stock of the 1st MTP joint (large bone cyst >1 cm, avascular necrosis)
* Allergy to polyvinyl alcohol
* Anyone unable to commit to follow up appointments
* Patients with significant medical comorbidities that make them unsuitable for elective surgery.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt M Rongstad, MD, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Madison
Locations (1):
- UW Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam A, Chan JJ, Surace MF, Vulcano E. Hallux rigidus: How do I approach it? World J Orthop. 2017 May 18;8(5):364-371. doi: 10.5312/wjo.v8.i5.364. eCollection 2017 May 18. PMID 28567339
- [Background] Baumhauer JF, Singh D, Glazebrook M, Blundell C, De Vries G, Le IL, Nielsen D, Pedersen ME, Sakellariou A, Solan M, Wansbrough G, Younger AS, Daniels T; for and on behalf of the CARTIVA Motion Study Group. Prospective, Randomized, Multi-centered Clinical Trial Assessing Safety and Efficacy of a Synthetic Cartilage Implant Versus First Metatarsophalangeal Arthrodesis in Advanced Hallux Rigidus. Foot Ankle Int. 2016 May;37(5):457-69. doi: 10.1177/1071100716635560. Epub 2016 Feb 27. PMID 26922669
- [Background] Nicolosi N, Hehemann C, Connors J, Boike A. Long-Term Follow-Up of the Cheilectomy for Degenerative Joint Disease of the First Metatarsophalangeal Joint. J Foot Ankle Surg. 2015 Nov-Dec;54(6):1010-20. doi: 10.1053/j.jfas.2014.12.035. Epub 2015 May 14. PMID 25981441
- [Background] Gould N, Schneider W, Ashikaga T. Epidemiological survey of foot problems in the continental United States: 1978-1979. Foot Ankle. 1980 Jul;1(1):8-10. doi: 10.1177/107110078000100104. PMID 6115797
- [Background] Lucas DE, Hunt KJ. Hallux Rigidus: Relevant Anatomy and Pathophysiology. Foot Ankle Clin. 2015 Sep;20(3):381-9. doi: 10.1016/j.fcl.2015.04.001. Epub 2015 Jul 4. PMID 26320553
- [Background] Kunnasegaran R, Thevendran G. Hallux Rigidus: Nonoperative Treatment and Orthotics. Foot Ankle Clin. 2015 Sep;20(3):401-12. doi: 10.1016/j.fcl.2015.04.003. Epub 2015 Jun 9. PMID 26320555
- [Background] Yee G, Lau J. Current concepts review: hallux rigidus. Foot Ankle Int. 2008 Jun;29(6):637-46. doi: 10.3113/FAI.2008.0637. No abstract available. PMID 18549766
- [Background] Coughlin MJ, Shurnas PS. Hallux rigidus. Grading and long-term results of operative treatment. J Bone Joint Surg Am. 2003 Nov;85(11):2072-88. PMID 14630834
- [Background] Sullivan MR. Hallux rigidus: MTP implant arthroplasty. Foot Ankle Clin. 2009 Mar;14(1):33-42. doi: 10.1016/j.fcl.2008.11.009. PMID 19232990
- [Background] Chee YH, Clement N, Ahmed I, Thomson CE, Gibson JN. Functional outcomes following ceramic total joint replacement for hallux rigidus. Foot Ankle Surg. 2011 Mar;17(1):8-12. doi: 10.1016/j.fas.2009.11.005. PMID 21276558
- [Background] Daniels TR, Younger AS, Penner MJ, Wing KJ, Miniaci-Coxhead SL, Pinsker E, Glazebrook M. Midterm Outcomes of Polyvinyl Alcohol Hydrogel Hemiarthroplasty of the First Metatarsophalangeal Joint in Advanced Hallux Rigidus. Foot Ankle Int. 2017 Mar;38(3):243-247. doi: 10.1177/1071100716679979. Epub 2016 Dec 7. PMID 27909032
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Madeley NJ, Wing KJ, Topliss C, Penner MJ, Glazebrook MA, Younger AS. Responsiveness and validity of the SF-36, Ankle Osteoarthritis Scale, AOFAS Ankle Hindfoot Score, and Foot Function Index in end stage ankle arthritis. Foot Ankle Int. 2012 Jan;33(1):57-63. doi: 10.3113/FAI.2012.0057. PMID 22381237
- [Background] Cullen B, Stern AL, Weinraub G. Rate of Revision After Cheilectomy Versus Decompression Osteotomy in Early-Stage Hallux Rigidus. J Foot Ankle Surg. 2017 May-Jun;56(3):586-588. doi: 10.1053/j.jfas.2017.01.038. PMID 28476391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2019 and September 2021, 20 participants were enrolled in the study and randomized. Surgical treatments began in July 2021.
Groups:
- Cartiva Hemiarthroplasty: Cartiva implant: The procedure starts with a small incision over the top of the 1st MTP joint. The joint is exposed. Bone spurs on the metatarsal and proximal phalanx are resected, leaving approximately 2 mm of surrounding bone on the metatarsal head. A guide pin is placed within the metatarsal and a drill is then used to create a site for the implant. The implant is then placed using the implant introducer. The incision is then closed and a sterile dressing is placed.
Period: Overall Study
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Started | 9 | 11
Completed Surgery | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Full Range); unit: years] | 62.1 [42 to 75] | 58.4 [50 to 72] | 60.25 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Number of Participants Who Smoke [Count of Participants; unit: Participants] | 0 | 1 | 1
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.5 [19.9 to 42.6] | 25.1 [20.1 to 32] | 26.5 [19.9 to 42.6]
Preoperative first metatarsophalangeal (MTP) peak active dorsiflexion (PAD) [Mean (Full Range); unit: degrees] | 30.0 [4.0 to 44.0] | 30.0 [20.0 to 50.0] | 30.0 [4.0 to 50.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Foot and Ankle Ability: Assessment by Foot and Ankle Ability Measure (FAAM-ADL) Questionnaire
Description: The Foot and Ankle Ability Measure (FAAM-ADL) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. The 21-item FAAM-ADL Questionnaire: scored as N/A, unable to do, extreme difficulty, moderate difficulty, slight difficulty, no difficulty, and/or a percentage (scale from 0-100, where higher scores indicate better physical function).
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
score on a scale
  Pre-operative: number analyzed (Participants) | 6 | 8
  Pre-operative | 77.5 (15.6) | 74 (19.3)
  post-operative week 2: number analyzed (Participants) | 1 | 1
  post-operative week 2 | 33 (NA) — data from 1 participant | 61 (NA) — data from 1 participant
  week 6: number analyzed (Participants) | 3 | 3
  week 6 | 71 (19.9) | 75 (15.5)
  month 3: number analyzed (Participants) | 6 | 5
  month 3 | 92 (5.1) | 92 (23.3)
  year 1: number analyzed (Participants) | 9 | 9
  year 1 | 89 (7.2) | 95 (20.3)
  year 2: number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Foot and Ankle Ability: Assessment by Foot and Ankle Ability Measure (FAAM-Sports) Questionnaire
Description: The Foot and Ankle Ability Measure (FAAM-Sports) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. FAAM-Sports Questionnaire is an 8-item survey: scored as N/A, unable to do, extreme difficulty, moderate difficulty, slight difficulty, no difficulty, and/or a percentage (scale from 0-100, where higher scores indicate higher level of physical function).
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
score on a scale
  pre-operative: number analyzed (Participants) | 6 | 8
  pre-operative | 68 (21.7) | 60.5 (29.7)
  post-operative week 2: number analyzed (Participants) | 1 | 1
  post-operative week 2 | 6 (NA) — data from 1 participant | 19 (NA) — data from 1 participant
  week 6: number analyzed (Participants) | 3 | 2
  week 6 | 18 (21.5) | 31.5 (13.4)
  month 3: number analyzed (Participants) | 5 | 5
  month 3 | 67 (24.3) | 78 (30.5)
  year 1: number analyzed (Participants) | 8 | 8
  year 1 | 67.5 (17.9) | 79 (28.8)
  year 2: number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Patient Health: Assessment by Short Form-36 Physical Component Scores (SF-36 PCS) Questionnaire
Description: The SF-36 is an indicator of overall health status. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability, higher scores = less disability
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
score on a scale
  Pre-operative: number analyzed (Participants) | 9 | 9
  Pre-operative | 35.5 (7.7) | 44.1 (10.4)
  post-operative week 2: number analyzed (Participants) | 3 | 3
  post-operative week 2 | 25.5 (12.1) | 33.5 (1.0)
  week 6: number analyzed (Participants) | 4 | 5
  week 6 | 32.7 (6.8) | 41.3 (10.6)
  month 3: number analyzed (Participants) | 5 | 4
  month 3 | 46.4 (3.6) | 54 (17.5)
  year 1: number analyzed (Participants) | 8 | 9
  year 1 | 50.4 (6.5) | 50.1 (11.1)
  year 2: number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Patient Health: Assessment by Short Form-36 Mental Component Scores (SF-36 MCS) Questionnaire
Description: as for outcome 3
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
score on a scale
  Pre-operative: number analyzed (Participants) | 9 | 8
  Pre-operative | 54.8 (5.1) | 58.2 (5.3)
  Post-operative week 2: number analyzed (Participants) | 3 | 3
  Post-operative week 2 | 55.8 (4.0) | 57.8 (16.6)
  week 6: number analyzed (Participants) | 4 | 4
  week 6 | 59.5 (3.0) | 58.65 (3.7)
  month 3: number analyzed (Participants) | 5 | 5
  month 3 | 55.8 (7.1) | 55.6 (8.7)
  year 1: number analyzed (Participants) | 9 | 9
  year 1 | 58.3 (4.1) | 58.2 (12)
  year 2: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in First MTP Peak Active Dorsiflexion
Description: This is a measure of the amount of dorsiflexion of the first metatarsophalangeal joint. It is performed by the clinician and measured with a protractor in clinic. It was measured preoperatively and post operatively.
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: degrees
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
degrees
  Pre-operative: number analyzed (Participants) | 8 | 7
  Pre-operative | 30 (8.8) | 30 (13.4)
  Post-operative week 2: number analyzed (Participants) | 2 | 3
  Post-operative week 2 | 33.5 (16.3) | 45 (8.7)
  6 weeks: number analyzed (Participants) | 4 | 5
  6 weeks | 33.5 (15.8) | 35 (12.4)
  3 months: number analyzed (Participants) | 2 | 4
  3 months | 47 (12.7) | 50 (21.4)
  year 1: number analyzed (Participants) | 5 | 5
  year 1 | 35 (14.3) | 45 (14)
  year 2: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change Visual Analog Scale (VAS) for Pain
Description: The VAS for pain is measured on a 0 to 100 point scale where 0 represents no pain and 100 indicates pain as bad as it could possibly be.
Time Frame: pre-operative baseline, post-operative Week 2, Week 6, Month 3, Year 1, and Year 2
Population: Study was terminated before the final time point per protocol.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
Number analyzed (Participants) | 9 | 10
score on a scale
  Pre-operative: number analyzed (Participants) | 8 | 7
  Pre-operative | 48 (20.7) | 56 (29.3)
  Post-operative week 2: number analyzed (Participants) | 1 | 1
  Post-operative week 2 | 40 (NA) — data from 1 participant | 75 (NA) — data from 1 participant
  week 6: number analyzed (Participants) | 3 | 2
  week 6 | 40 (36) | 30 (35.4)
  month 3: number analyzed (Participants) | 5 | 5
  month 3 | 7 (6.1) | 10 (32.7)
  year 1: number analyzed (Participants) | 7 | 9
  year 1 | 17 (13.4) | 2 (17.6)
  year 2: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1.5 years
Arm/Group | Cartiva Hemiarthroplasty | Cheilectomy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cartiva Hemiarthroplasty (N=9) | Cheilectomy (N=10)
Wound Dehiscence (Infections and infestations) | 0 (0) | 1 (1) — post-operative wound dehiscence which was treated with local wound cares and oral antibiotics
Pain (General disorders) | 1 (1) | 1 (1) — 1 participant in the cartiva group underwent a steroid injection for pain 6 months post operatively. In the cheilectomy group, 1 participant underwent a steroid injection for pain 3 months post operatively.
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1) — revision surgery with conversion of cheilectomy to a 1st MTP arthrodesis approximately 1.5 years after the index procedure

LIMITATIONS AND CAVEATS:
This study was terminated early and was not powered for meaningful results per the protocol. Median data at each timepoint are reported here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03935880/Prot_SAP_000.pdf